CLINICAL TRIAL: NCT06505330
Title: Study of the Effects of Probiotics on the Upper Respiratory Tract Microbiome and the Prevention of Otitis Media With Effusion in Children With Cleft Palate
Brief Title: Respiratory Tract Microbiome and Probiotics in Children With Cleft Palate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B3002024000099
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Otitis Media in Children; Cleft Palate Children
Keywords: otitis media; upper respiratory tract microbiome; cleft palate; probiotics; Lacticaseibacillus rhamnosus GG
MeSH Terms: conditions — Otitis Media; Cleft Palate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention)
- Probiotic group (Experimental): Dietary Supplement: Probactiol Mini 6 droplets of Probactiol Baby contain 1 billion bacteria (Lactobacillus rhamnosus GG and Bifidobacterium lactis BB-12)
  Interventions: Dietary Supplement: Probactiol Baby

INTERVENTIONS:
Dietary Supplement: Probactiol Baby — Dietary Supplement: Probactiol Mini 6 droplets of Probactiol Mini daily intake for 13 months
  Arms: Probiotic group

SUMMARY:
Otitis media with effusion (OME) involves fluid accumulation in the middle ear without infection, sometimes causing discomfort and hearing loss in children. Persistent middle ear fluid lasting over 3 months may require treatment, including placement of ventilation tubes if it affects hearing.

Children with a cleft palate are at higher risk for otorrea after ventilation tube placement. Treatment typically involves antibiotic drops and ear cleaning by an ENT doctor, often requiring repeated visits, which may impact quality of life for both the child and the parents.

The mouth, throat, and nose harbor bacteria that can influence ear infections. This study aims to determine if probiotics can alter the bacteria in the nasopharynx and middle ear fluid and reduce the number of episodes of eardischarge following ventilation tube placement in children with cleft palate.

Using Lacticaseibacillus rhamnosus GG and Bifidobacterium lactis BB-12 from Bactiol® Baby (Metagenics), patients will be divided into two groups: one receiving probiotic drops and one not. The study will assess if probiotics can reduce the number of episodes with ear discharge in children with cleft palate, by examining the following:

1. The airway microbiome composition in children with cleft palates.
2. Whether oral probiotics can reduce the number and duration of ear discharge episodes.

ELIGIBILITY:
Inclusion Criteria:

* cleft palate & lip (uni/bilateral) or cleft palate
* No syndromal disorders

Exclusion Criteria:

* syndromal disorder
* history of ventilation tube placement

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2028-06-24 (Estimated)

PRIMARY OUTCOMES:
Microbiome composition | over the study period (= 13 months)
  Longitudinal study of the composition of the URT microbiome (alpha, beta diversity and individual taxa), more specific the oral cavity, rhinopharynx, and middle ears. Analysis will be done with 16S amplicon sequencing or shotgun sequencing.
Number of episodes of otorrea | over the study period (= 13 months)
  Document the number and duration of episodes of otorrea after ventilation tube placement

SECONDARY OUTCOMES:
Effect of probiotics on the composition of the URT microbiome | over the study period (= 13 months)
  Longitudinal study of the effect of probiotics on the composition of the upper respiratory tract microbiome in children with cleft palate. This will be analysed by 16S amplicon sequencing or shotgun sequencing, and qPCR.
Transfer of bacteria | over the study period (= 13 months)
  Follow-up of the transfer of orally administered probiotic bacteria to the upper respiratory tract (rhinopharynx, middle ears, oral cavity). Done with qPCR
Differences in abundances of lactic acid bacteria in control/probiotic treatment group | over the study period (= 13 months)
  Analysis of the differences in abundances of lactic acid bacteria in the microbiome of patients with cleft palate with/without the administration of probiotics, done by sequencing and qPCR

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No